CLINICAL TRIAL: NCT07405021
Title: Effect of Vagus Nerve Stimulation on Pain Intensity, Nerve Conduction Studies and Functional Outcomes in Diabetic Peripheral Neuropathy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Mamdouh Nematallah, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005474
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Transcutaneous Vagal Nerve Stimulation (tVNS); Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Vagus nerve stimulation (Experimental): Patients will receive the same traditional physical therapy as in traditional physical therapy group in addition to 30 min of transcutaneous auricular vagus nerve stimulation 5 sessions per week for 6 weeks.
  Interventions: Other: Conventional physical therapy program; Device: Transcutaneous auricular vagus nerve stimulation
- traditional physical therapy (Active Comparator): Patients will receive 30 min of traditional physical therapy, and 30 min of placebo Non-Invasive vagus nerve stimulation, 5 sessions per week for 6 weeks
  Interventions: Other: Conventional physical therapy program; Device: Sham therapy

INTERVENTIONS:
Other: Conventional physical therapy program — Flexibility exercises:
  Gentle passive progressive stretching and self-stretches for lower limbs selected muscles.
  Muscle strengthening (using a variety of modes as appropriate e.g. isometric, graded weight progression, open and close chain) Aerobic activity. Posture and balance training (for falls prevention and stability). Gait (can improve proprioception and gait pattern in patients with diabetic neuropathy
Device: Sham therapy — A sterile cotton ball will be placed in the ear after sterilizing the cavum conchae and cymba conchae with 75% alcohol. The stimulation electrode will be inserted into the cotton ball, and then the cotton ball will be fixed after ensuring that the stimulator does not touch the skin; the lead wire will be connected. The therapeutic apparatus will be turned on, and the parameters will be the same as those for the transcutaneous vagus nerve stimulation group. All patients will see the lights flashing when the stimulator is running
  Arms: traditional physical therapy
Device: Transcutaneous auricular vagus nerve stimulation — The antihelix and cymba concha will be sterilized with 75% alcohol, and then the nerve stimulation electrode (the ear clips) will be attached. The positive pole of the lead will be connected to the antihelix, and the negative pole will be connected to the cymba concha The device parameters include a wave width of 0.2 ms ± 30% and a pulse frequency of 20 Hz. Current intensity will gradually increase to a tolerable level of 4-6 mA, with stimulation lasting for 30 minutes. Heart rates of participants will be monitored continuously, with stimulation ceasing if rates drop below 50 beats per minute. Both the study and control groups will receive the same conventional physical therapy program.
  Arms: Transcutaneous Vagus nerve stimulation

SUMMARY:
To evaluate the efficacy of vagus nerve stimulation in reducing neuropathic pain, symptom severity, electrophysiological studies and functional outcomes in patients with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Diabetes is a major global health problem affecting half a billion people worldwide. Its global prevalence is rising at an alarming rate and has been forecast to reach 700 million by 2045. Diabetic neuropathy is an important and common complication of diabetes, with a lifetime prevalence of more than 50% among people with diabetes. Diabetic neuropathy is an insidious and often disabling disease.

Sensory symptoms are diverse, ranging from numbness to dysesthesia, pain and allodynia, and typically begin in the feet and spread proximally. Motor function can also be affected, preventing patients from engaging in activities of daily living. More recently, the considerable psychosocial and quality of life impacts of Diabetic neuropathy have been recognized. Furthermore, Diabetic neuropathy is a major risk factor for diabetic foot ulceration, which is an independent risk factor for lower limb amputation and mortality. The associated economic burden is high; the annual cost of managing Diabetic neuropathy exceeds billions of dollars in different countries .

Current treatments are purely symptomatic and the most commonly recommended first-line agents include anticonvulsants (gabapentin and pregabalin), serotonin-noradrenaline reuptake inhibitors, and tricyclic antidepressants. Unfortunately, the therapeutic effect may offset by intolerable adverse effects.

In this study, evidence for a potentially effective, non-pharmacological treatment option for Diabetic neuropathy will be provided. Positive findings could lead to improved management strategies for Diabetic neuropathy, reducing the burden of chronic pain and enhancing the overall well-being of diabetic patients. Vagus nerve stimulation has emerged as a potential intervention, offering promise in modulating neuropathic pain and improving functional outcomes.

Furthermore, understanding the mechanisms through which transcutaneous Vagus nerve stimulation affects pain and nerve function may offer insights into broader applications of vagus nerve stimulation in other neuropathic conditions. This research could pave the way for future studies and clinical applications, positioning transcutaneous Vagus nerve stimulation as a valuable tool in the multidisciplinary approach to managing diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria

* Thirty patients diagnosed with diabetic neuropathy of both genders.
* Age range between 45 and 60 years.
* Presence of numbness and/or pain in the feet with no other identifiable cause.
* Pain characterized as stabbing, electric shock-like, or burning in nature.
* Presence of glove-stocking sensory changes and abnormal sensations in the distal lower limbs.
* Ability to ambulate independently without assistance.
* Patients under full medical control.
* Hemoglobin A1c levels ranging from 6.5% to 7%.
* History of diabetes mellitus for more than 5 years.

Exclusion Criteria

* Implantation of cardiac pacemakers or other electrical stimulation devices.
* Presence of sinus bradycardia, sick sinus syndrome, or other cardiac arrhythmias.
* Lumbar radiculopathy.
* Psychiatric or mental disorders or history of seizures.
* Visual or auditory impairments or tremors affecting balance.
* Presence of other neuromuscular disorders.
* Foot deformities or active foot ulcers.
* History of lower limb surgical operations.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity | at baseline and after 6 weeks.
  The Neuropathic Pain Questionnaire-Short Form consists of 3 items assessing tingling pain, numbness, and increased pain due to touch. Patients rate each item on a scale from 0 (no pain) to 100 (worst imaginable pain/greatest intensity). translated version of Neuropathic Pain Questionnaire-Short Form is reliable and valid for use, to evaluate and diagnose neuropathic pain among Arabic-speaking patients

SECONDARY OUTCOMES:
assessment of sensory nerve action optential. | at baseline and after 6 weeks.
  nerve conduction studies is one of the gold standard techniques for diagnosing diabetic poly neuropathy Neuropack Nihon Kohden, Model MEB- 9400, Serial number:00218. (Figure The device is used for electrodiagnosis of diabetic peripheral neuropathy. It is used to measure the sensory nerve action optential.
assessment of sensory nerve conduction velocity of lower limb | at baseline and after 6 weeks.
  nerve conduction studies is one of the gold standard techniques for diagnosing diabetic poly neuropathy Neuropack Nihon Kohden, Model MEB- 9400, Serial number:00218. (Figure The device is used for electrodiagnosis of diabetic peripheral neuropathy. It is used to measure the Sensory conduction velocity
assessment of Sensory distal latency of lower limb | at baseline and after 6 weeks.
  nerve conduction studies is one of the gold standard techniques for diagnosing diabetic poly neuropathy Neuropack Nihon Kohden, Model MEB- 9400, Serial number:00218. (Figure The device is used for electrodiagnosis of diabetic peripheral neuropathy. It is used to measure the Sensory distal latency
assessment of lower limb functional scale | at baseline and after 6 weeks.
  is a widely used patient-reported questionnaire with 20 items to assess difficulty with daily activities due to lower limb problems, scoring from 0 (extreme difficulty) to 4 (no difficulty) for each item, totaling 0-80 points, with higher scores indicating better function.
assessment of motor nerve conduction velocity of lower limb | at baseline and after 6 weeks.
  nerve conduction studies is one of the gold standard techniques for diagnosing diabetic poly neuropathy Neuropack Nihon Kohden, Model MEB- 9400, Serial number:00218. (Figure The device is used for electrodiagnosis of diabetic peripheral neuropathy. It is used to measure the motor conduction velocity.
assessment of motor distal latency | at baseline and after 6 weeks.
  nerve conduction studies is one of the gold standard techniques for diagnosing diabetic poly neuropathy Neuropack Nihon Kohden, Model MEB- 9400, Serial number:00218. (Figure The device is used for electrodiagnosis of diabetic peripheral neuropathy. It is used to measure the motor distal latency
assessment of motor nerve action optential. | at baseline and after 6 weeks.
  nerve conduction studies is one of the gold standard techniques for diagnosing diabetic poly neuropathy Neuropack Nihon Kohden, Model MEB- 9400, Serial number:00218. (Figure The device is used for electrodiagnosis of diabetic peripheral neuropathy. It is used to measure the motor nerve action optential.

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic, faculty of physical therapy, Horus university, Damietta, Egypt